CLINICAL TRIAL: NCT00516828
Title: A Phase I/II Study of Sorafenib (BAY 43-9006) in Combination With Low Dose ARA-C (CYTARABINE) in Elderly Patients With AML or High-Risk MDS
Brief Title: Sorafenib and Low Dose Cytarabine in Older Patients With Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I186; CAN-NCIC-IND186 (Registry Identifier: NCI US - Physician Data Query); CDR0000560975 (Other: PDQ)
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Congenital Abnormalities | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sorafenib and Cytarabine (Experimental): Cytarabine: subcutaneously twice daily from day 1 - 10. Sorafenib: Days 2-28; at the dose level assigned at registration. Sorafenib will be given orally twice daily.
  Interventions: Drug: cytarabine

INTERVENTIONS:
Drug: cytarabine — subcutaneously twice daily from Day 1 to 10

SUMMARY:
RATIONALE: Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the cancer. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with cytarabine may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving sorafenib together with cytarabine and to see how well it works in treating older patients with acute myeloid leukemia or high-risk myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the recommended dose of sorafenib tosylate and cytarabine when given in combination to elderly patients with acute myeloid leukemia or high-risk myelodysplastic syndromes who are not suitable for intensive chemotherapy. (Phase I)
* To determine the safety, tolerability, toxicity profile, and dose-limiting toxicities in patients treated with this regimen. (Phase I)
* To estimate the efficacy (as measured by complete response rate) in patients treated with this regimen. (Phase II)
* To describe the toxic effects and overall response rate (complete and partial) in patients treated with this regimen. (Phase II)
* To evaluate potential correlates of response in translational research studies including FLT-3 internal tandem duplications and point mutations in blasts. (Phase II)

OUTLINE: This is a multicenter study.

* Phase I: Patients receive oral sorafenib tosylate twice daily on days 2-28 and cytarabine subcutaneously twice daily on days 1-10 at the dose level assigned at registration. Doses of both drugs will be escalated and the recommended doses for the combination will be determined. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who respond to treatment will receive 2 cycles after response criteria are met.
* Phase II: Patients receive sorafenib tosylate and cytarabine as in phase I at the recommended doses for the combination determined in phase I.

Bone marrow (or blood) samples are collected at baseline and at the end of each course of study treatment. Baseline samples are analyzed for mutational status of FLT-3 (i.e., internal tandem duplication [ITD] and point mutations).

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter until progression and toxicities resolve.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML) by FAB criteria (By morphology and routine histochemistry and confirmed, when possible, by flow cytometric analysis of surface immunophenotype; co-expression of lymphoid markers permitted)
  * High-risk myelodysplastic syndromes defined as IPSS category of intermediate-2 or greater
* Must be considered unsuitable for intensive chemotherapy regimens
* No documented CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* AST and ALT ≤ 2 times upper limit of normal (ULN)
* Bilirubin normal
* Creatinine ≤ 1.2 times ULN OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of other malignancies, except adequately treated nonmelanoma skin cancer, curatively treated in situ carcinoma of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* No upper gastrointestinal or other conditions that would preclude compliance with or administration of oral medication
* No serious illness or medical condition that would not permit the patient to be managed according to the protocol, including any of the following:

  * History of significant neurologic or psychiatric disorder that would impair the ability to obtain consent
  * Active, uncontrolled, serious infections
  * Active peptic ulcer disease
  * Evidence of bleeding diathesis
* No myocardial infarction within the past 6 months
* No congestive heart failure
* No unstable angina
* No active cardiomyopathy or unstable ventricular arrhythmia
* No poorly controlled hypertension (e.g., systolic BP ≥ 150 mm Hg or diastolic BP ≥ 95 mm Hg)
* No known hypersensitivity to the study drugs or their components
* No preexisting hypothyroidism prior to enrollment unless patient is euthyroid on medication
* No neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* At least 2 days since prior hydroxyurea
* No other prior chemotherapy
* No concurrent therapeutic doses (≥ 2 mg/day) of anticoagulants (e.g., warfarin)

  * Doses of up to 2 mg/day given for prophylaxis of thrombosis are accepted provided INR is ≤ 1.5
* No other concurrent experimental drugs or anticancer therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-11-27 (Actual); Primary Completion 2010-03-18 (Actual); Study Completion 2013-01-10 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of sorafenib tosylate when given in combination with cytarabine (Phase I) | 29 months
Dose-limiting toxicity (Phase I) | 29 months
Complete remission (Phase II) | 29 months

SECONDARY OUTCOMES:
Overall response rate (complete and partial response) (Phase II) | 29 months
Time to progression (Phase II) | 29 months
Overall survival (Phase II) | 29 months
FLT-3 ITD endpoint mutation response correlation. | 29 months
Toxicity (Phase II) | 29 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Leber, MD, FRCPC, Study Chair — McMaster Children's Hospital at Hamilton Health Sciences; David A. MacDonald, MD, Study Chair — Nova Scotia Cancer Centre
Locations (4):
- Canada (4):
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Macdonal DA, Assouline SE, Brandwein J, Kamel-Reid S, Eisenhauer EA, Couban S, Foo A, Leber B. Phase I/II study of low-dose cytarabine with sorafenib as first-line therapy of elderly patients with AML or high-risk myelodysplastic syndrome. J Clin Oncology 28[15s, abstr 6564]. 2010.